CLINICAL TRIAL: NCT05229510
Title: A Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Inhaled Virazole Administered Via Air-Jet Nebulizer in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of Inhaled Virazole Administered Via Air-Jet Nebulizer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BHC-RIB-5101
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- 50 mg/mL Virazole (10 ml total volume) (Experimental): 50 mg/mL Virazole (10 ml total volume) aerosolized and administered until solution depleted (approximate time of treatment is 20 minutes).
  Interventions: Drug: 50 mg/mL Virazole Inhalant Product
- 50 mg/mL Virazole (20 ml total volume) (Experimental): 50 mg/mL Virazole (20 ml total volume) aerosolized and administered until solution depleted (approximate time of treatment is 40 minutes).
  Interventions: Drug: 50 mg/mL Virazole Inhalant Product
- 100 mg/mL Virazole (10 ml total volume) (Experimental): 100 mg/mL Virazole (10 ml total volume) aerosolized and administered until solution depleted (approximate time of treatment is 20 minutes).
  Interventions: Drug: 100 mg/mL Virazole Inhalant Product
- 100 mg/mL Virazole (20 ml total volume) (Experimental): 100 mg/mL Virazole (20 ml total volume) aerosolized and administered until solution depleted (approximate time of treatment is 40 minutes).
  Interventions: Drug: 100 mg/mL Virazole Inhalant Product
- Placebo (Placebo Comparator): Placebo aerosolized and administered until solution depleted
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50 mg/mL Virazole Inhalant Product — 50 mg/mL Virazole (10 or 20 ml total volume) aerosolized and administered until solution depleted
  Arms: 50 mg/mL Virazole (10 ml total volume); 50 mg/mL Virazole (20 ml total volume)
Drug: 100 mg/mL Virazole Inhalant Product — 100 mg/mL Virazole (10 or 20 ml total volume) aerosolized and administered until solution depleted
  Arms: 100 mg/mL Virazole (10 ml total volume); 100 mg/mL Virazole (20 ml total volume)
Drug: Placebo — Placebo (10 or 20 ml total volume) aerosolized and administered until solution depleted
  Arms: Placebo

SUMMARY:
This study is a Phase 1a, randomized, double-blind, placebo-controlled, safety, tolerability, and PK study in healthy adult volunteers.

Participants were screened for eligibility within 14 days prior to enrollment. Four successive cohorts were enrolled, with each cohort receiving a single dose of Virazole or placebo using different delivery regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female ≥ 18 and ≤65 years of age.
2. For a female, must be of non-childbearing potential according to 1 of the following criteria at least 6 months prior to screening:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * post-menopausal with spontaneous amenorrhea for ≥ 12 consecutive months with follicle-stimulating hormone [FSH] > 25.8 mIU/mL; or
   * having had bilateral oophorectomy (with or without hysterectomy).
3. For a male subject must be vasectomized with confirmed postvasectomy semen analysis or a male subject with a documented diagnostic of infertility.
4. Subject willing and able to provide written informed consent.
5. Subject has a body mass index (BMI) ≥ 18.50 and < 30.00 kg/m2.
6. Subject is in good general health without clinically significant haematological, cardiac, respiratory, renal, endocrine, gastrointestinal, psychiatric, hepatic, or malignant disease, as determined by the Investigator.
7. Subject has suitable venous access for blood sampling

Exclusion Criteria:

1. Subject has a history of hypersensitivity to ribavirin.
2. Subject has a history of asthma, COPD, or bronchospasm.
3. Subject has anemia defined as hemoglobin or RBC <75% of the institutional lower limit of normal for age and gender.
4. Subject has any major illness or systemic infection (including COVID-19) within 4 weeks of the Screening Visit or has a clinically relevant history or is currently suffering from a disease or condition that, in the opinion of the Investigator, may affect the evaluation of the study drug or place the subjects at undue risk.
5. Subject is seropositive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV), or positive for SARS-CoV-2 at Screening.
6. Subject has a clinically relevant history of or current evidence of abuse of alcohol or other drug(s).
7. Subject is currently a tobacco smoker or was a tobacco smoker within 6 months of the Baseline Visit.
8. Subject has donated 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, Clinical Studies, etc.) in the previous 56 days prior to the Baseline Visit.
9. Subject is currently participating in any drug or device clinical investigation or has received an investigational agent or approved drug that, in the Investigator's judgement, may have a chemical or pharmacological interaction with Virazole if administered within 5 half-lives or 30 days of the Baseline Visit.
10. Subject has any condition that could cause noncompliance with treatment or may otherwise contraindicate the subject's participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Bausch Site 1, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No